CLINICAL TRIAL: NCT07105267
Title: A Proof of Concept Study : Open Label Phase IIa Trial Evaluating the Effect and Safety of Transplantation of Fecal Microbiota in Children With Autism Spectrum Disorders and Gastrointestinal Symptoms
Brief Title: Open Label Phase IIa Trial Evaluating the Effect and Safety of Transplantation of Fecal Microbiota in Children With Autism Spectrum Disorders and Gastrointestinal Symptoms
Acronym: FELICITA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation initiative autisme (Unknown); Fondation Erie (Unknown); Biocodex microbiota fondation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP241418; 2025-520539-17-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-21; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder; Fecal Microbiota Transplantation (FMT)
Keywords: Austim Spectrum Disorder; FMT; gastrointestinal symptom,
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — FMT protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Felictia Arm (Experimental): FMT
  Interventions: Drug: FMT Protocol

INTERVENTIONS:
Drug: FMT Protocol — FMT protocol Samples (urine, blood, stool) collection Psychological examination Pediatric quality of life Scale Bristol Stool form Scale

SUMMARY:
Autism Spectrum Disorders (ASD), affect approximately 1% of the general population and are characterized by impairments in social communication associated with repetitive/stereotyped behaviors. Approximately one-third of these patients display gastrointestinal (GI) symptoms, and a growing number of studies suggest abnormalities of gut microbiota in ASD. Gut microbiota and the brain interact through complex pathways. Preliminary evidence in adults with ASD suggests that modulation of the gut microbiota by probiotics and/or prebiotics and more recently by fecal microbiota transplantation could improve GI symptoms but also socio-communication deficit, with persistent improvement at year 2.

DETAILED DESCRIPTION:
1. Screening :

   Screening will be done in ASD units of child psychiatry departments of Robert Debré
2. Information of patients and their families Information will be delivered in the child psychiatry department of Robert Debré hospital.
3. Inclusion Consent will be collected in CIC of Robert Debré hospital during the initial visit by child psychiatrist 7 to 15 days after information from the patient's family.
4. Patient follow-up during trial Initial visit: for parents and patient information. Further visits (W4, W18, W24, M12): treatment administrations will be done at the CIC. Subjects will be evaluated on efficacy and safety and acceptability. Stool, urine and blood samples will be collected.

   Phone visits (W11 and M9): Safety and the Acceptability questionnaire (parents) will be evaluated.
5. Products: donor and transplant preparation
6. Same administration schedule in FMT

   * D1 to D4: Vancomycin (10mg/kg, 4 times a day). 1st dose in the CIC, the 3 others at home
   * D4: Picoprep® treatment at home
   * D5: First FMT using rectal enema (100ml = 25g of stool from donor) using Foley probe (rectal administration) in CIC
   * D12: Second FMT using rectal enema (100ml = 25g of stool from donor) using Foley probe (rectal administration) in CIC
   * D19: Third FMT using rectal enema (100ml = 25g of stool from donor) using Foley probe (rectal administration) in CIC

ELIGIBILITY:
Inclusion Criteria:

* ASD diagnosis based on DSM-5 criteria
* Gastrointestinal symptoms: at least a score of 5 on 1 of the 5 GSRS domains (diarrhea, abdominal pain, constipation, indigestion, reflux) for over a period of 1 year or more
* Age between 36 and 72 months
* Consent from all legal guardians
* Social insurance affiliation

Exclusion Criteria:

* Severe intellectual deficit (IQ<30) or another uncontrolled comorbidity (e.g. epilepsy)
* Recent change in ASD global care (cognitive behavioral therapy 6 weeks before inclusion)
* Actual or past psychotropic medication
* Contraindications to colon preparation (Picoprep®) and/or to Meopa)
* Severe or uncontrolled gastrointestinal symptoms (e.g. urgent treatment needed)
* Undernutrition (age related BMI < 3rd percentile)
* Inflammatory bowel disease
* Exclusive diet (gluten- or sugar-free)
* Rectal enema contraindication
* Antibiotic or antifungal therapy 3 months before inclusion
* Probiotics 2 months before inclusion or FMT 12 months before inclusion
* Vancomycin or Picoprep® or Meopa (including excipients) known allergy or intolerance Experimental therapeutic trial participation 3 months before inclusion

Ages: 36 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Score of the Gastrointestinal Symptoms Rating Scale (GSRS) | Week 18
  Assess initial efficacy on gastrointestinal (GI) symptoms of fecal microbiota transplantation (FMT) in children (36 to 72 months) with autism spectrum disorders (ASD (FMT) The Gastrointestinal Symptoms Rating Scale (GSRS) uses 15 items rated on a 7-point scale to assess gastrointestinal symptom severity, with total scores ranging from 15 (no symptoms) to 105 (very severe symptoms). Higher GSRS scores indicate more severe symptoms and a worse gastrointestinal outcome.

SECONDARY OUTCOMES:
Score of Vineland Adaptative Behavior Composite 3 scale | Day 0, Week 4, Week 18, Week 24, Month 12
  Estimate the effect of FMT on autistic core symptoms and global functioning (socio adaptivecapacities, social cognition, repetitive and stereotyped behaviors) The Vineland Adaptive Behavior Scales (VABS) standard scores for each domain and the overall Adaptive Behavior Composite (ABC) range from 20 (minimum) to 160 (maximum), with a mean of 100 and a standard deviation of 15. Higher Vineland scores indicate better adaptive functioning and more positive outcomes, whereas lower scores reflect greater impairment in adaptive behavior
Score of Pediatric Adverse Event Rating Scale | Day 0, Day 5, Week 4, Week 18, Week 24, Month 12
  FMT side effects (antibiotic therapy, GM transplantation from a healthy donor): Pediatric Adverse Event Rating Scale [evaluated by the investigator at day (D) 0, D5, W4, W18, W24, M12The Pediatric Adverse Event Rating Scale (PAERS) uses a combined score for each symptom that ranges from 0 (no symptom) to 5 (most severe/extreme symptom with impairment), based on symptom presence, functional impairment, and severity. Higher PAERS scores indicate more severe or impactful adverse events, representing a worse outcome]
Tolerability: Score of bristol Stool form | Day 0, Week 4, Week 18, Week 24, Month12
  Estimate FMT tolerability: completion of the FMT process and acceptability questionnaire (parents)
Score of Pediatric Quality of Life Inventory | Day 0, Week 18, Month 12
  Estimate FMT impact on children and parent's quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ELLUL, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debré Hospital, Paris, Ap-hp / DRCI, France